CLINICAL TRIAL: NCT00605956
Title: An Evaluation of the Photoallergy Potential of NatrOVA Creme Rinse - 1% in Healthy Volunteers
Brief Title: NatrOVA Photoallergy Study - NatrOVA Creme Rinse in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ParaPRO LLC (Industry)
Responsible Party: William C. Culpepper III, ParaPRO, LLC
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPN-108-08; HTR Study #07-128385-111
Record Dates: First submitted 2008-01-21; First posted 2008-02-01 (Estimated); Last update posted 2008-08-04 (Estimated); Status verified 2008-05

CONDITIONS: Head Lice
Keywords: head lice; NatrOVA Creme Rinse - 1% is intended for the treatment of head lice

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): NatrOVA Creme Rinse - 1% Spinosad
  Interventions: Drug: NatrOVA Creme Rinse - 1%
- 2 (Experimental): NatrOVA Vehicle - no Spinosad
  Interventions: Drug: NatrOVA Creme Rinse Vehicle Only
- 3 (Placebo Comparator): Blank Patch
  Interventions: Drug: Blank Patch

INTERVENTIONS:
Drug: NatrOVA Creme Rinse - 1% — NatrOVA Creme Rinse - 1% spinosad
  Arms: 1
Drug: NatrOVA Creme Rinse Vehicle Only — NatrOVA Creme Rinse Vehicle - no spinosad
  Arms: 2
Drug: Blank Patch — Blank Patch
  Arms: 3

SUMMARY:
Photoallergic reactions are assumed to be due to a delayed cell-mediated hypersensitivity response that requires the presence of ultraviolet irradiation. The predictive procedure is, therefore, based on modification of the Repeated Insult Patch Test (Kaidbey, 1991). Duplicate sets of patches of test articles are used with exposure of only one set to UV radiation and subsequent evaluation of both sets for skin reactions in order to compare irradiated versus non-irradiated test sites.

DETAILED DESCRIPTION:
The study consists of of following phases: screening, induction, rest, challenge, and re-challenge (if necessary). The study will be conducted as a randomized, evaluator-blind test design.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 18-65 years of age
* Has the ability to understand and has signed a written informed consent form and HIPAA authorization
* Females of childbearing potential must agree to use an adequate birth control
* Fitzpatrick (1988) skin type I, II, or III.

Exclusion Criteria:

* History of severe reactions from exposure to sunlight
* Known allergies or sensitivities to adhesives in patches, medical tape, or ingredients found in the test articles
* Inability to evaluate the skin in and around the test sites
* Diabetes requiring medication
* Clinical significant skin diseases which may contraindicate participation
* Asthma or any other severe respiratory disease requiring chronic medication
* Known immunological disorders such as HIV, AIDS, SLE and/or RA
* History, within the last six months, of current cancer, including skin cancer
* Mastectomy for cancer removal of lymph nodes draining test sites
* Epilepsy
* Pregnancy, lactation, or planning a pregnancy during the test period
* Chronic use of systemic antihistamine medication, or use within 14 days prior to Screening Visit
* Use of anti-inflammatory drugs (exception: acetaminophen and < 81 mg.day aspirin are permitted) within 2 days of Screening Visit
* Currently receiving allergy injections
* Currently taking or expecting to take any photosensitizing medications
* Use of immunosuppressive drugs
* Topical drugs used at the test sites within the last 7 days prior to screening
* Current participation in any clinical trial
* Participation in any patch test for irritation or sensitization or any test involving UV exposures within 4 wees of study start
* Use of any investigational therapy within the past 4 weeks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Visual grading of test site and assessments of adverse experiences | Evaluations over a 6 week period

CONTACTS AND LOCATIONS:
Overall Officials: John V. Murray, MD, Principal Investigator — Hill Top Research
Locations (1):
- Hill Top Research, St. Petersburg, Florida, United States

REFERENCES:
- See also: sponsor website — http://www.parapro.com